CLINICAL TRIAL: NCT02308410
Title: Effect of Tourniquet Application on Postoperative Functional Outcome Following Total Knee Arthroplasty; a Prospective Cohort Study
Brief Title: Effect of Tourniquet Application on Postoperative Functional Outcome Following Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Medicort Sports & Orthopedic Care (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Sponsor
Other Study IDs: Medicort Bergman Tourniquet
Record Dates: First submitted 2014-11-20; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
Keywords: Tourniquet; Postoperative outcome; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tourniquet group: This group received a pneumatic tourniquet during total knee arthroplasty.
  Interventions: Procedure: Tourniquet application during surgery
- Non-tourniquet group: This group received no tourniquet during total knee arthroplasty.

INTERVENTIONS:
Procedure: Tourniquet application during surgery — Both groups received usual care according to the orthopedic surgeons surgical preferences. One group received no tourniquet during surgery (non-tourniquet group) and the other group received a pneumatic tourniquet during surgery (tourniquet-group).
  Groups: Tourniquet group

SUMMARY:
A pneumatic tourniquet is often used during total knee arthroplasty. However, its effect on postoperative outcomes as soft tissue damage resulting in delayed recovery remains unclear. The purpose of the present study was to compare tourniquet use versus non-tourniquet use during total knee arthroplasty for short-term functional recovery.

DETAILED DESCRIPTION:
In a prospective cohort design, consecutive series of patients who underwent primary unilateral total knee arthroplasty (TKA) in the Bergman Clinic, the Netherlands were investigated. Patients scheduled for primary TKA due to osteoarthritis, age between 50 and 75 years and with Dutch language proficiency were eligible for inclusion. Exclusion criteria were inflammatory arthritis, severe cardiac complaints, severe pulmonary disorders, Body Mass Index (BMI) >35, severe coagulation disorders or hospitalization in the previous two months before surgery. Each patient included in the study signed informed consent. The research protocol was approved by the Regional Ethics Committee VCMO in Nieuwegein, the Netherlands, registration number W13.022.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled TKA due to osteoarthritis
* Age between 50 and 75 years
* Dutch language proficiency
* Signed informed consent

Exclusion Criteria:

* Inflammatory arthritis
* Severe cardiac complaints
* Severe pulmonary disorders
* Body Mass Index >35
* Severe coagulation disorders
* Hospitalization in the previous two months before surgery

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a prospective cohort design, consecutive series of patients who underwent primary unilateral total knee arthroplasty in the Bergman Clinic Naarden, the Netherlands were investigated.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Score (KOOS) questionnaire | 8 weeks
  The KOOS questionnaire was used to assess the functional outcome. Changes were evaluated from baseline at 8 weeks.

SECONDARY OUTCOMES:
Range of Motion (ROM) | Baseline, day 1, day 2, day 3 and 8 weeks
  A standard clinical 30cm goniometer was used to evaluated the ROM
Isometric bilateral strength | Baseline and 8 weeks
  Bilateral isometric strength of the lower limb was measured using hand-held dynamometry (HHD)
VAS questionnaire. | Baseline, day 1, day 2, day 3 and 8 weeks
  A 100mm Visual Analogue Scale was used for measuring current, minimal and maximal pain.
EQ-5D questionnaire | Baseline, day 1, day 2, day 3 and 8 weeks
  Quality of life was using the EQ05D questionnaire.

OTHER OUTCOMES:
Length of Stay (LOS) | Baseline, day 1, day 2 and day 3
  The total length of each the patients in hospital stay was calculated and evaluated for comparison between both groups.
Used analgesics | Baseline, day 1, day 2 and day 3
  During the clinical phase, analgesic use was noted whereas the doses and time interval of each medication was recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Bergman Clinic Naarden, Naarden, North Holland
  - Medicort Sports & Orthopedic Care, Naarden, North Holland

REFERENCES:
- [Result] Ejaz A, Laursen AC, Kappel A, Laursen MB, Jakobsen T, Rasmussen S, Nielsen PT. Faster recovery without the use of a tourniquet in total knee arthroplasty. Acta Orthop. 2014 Aug;85(4):422-6. doi: 10.3109/17453674.2014.931197. Epub 2014 Jun 23. PMID 24954487